CLINICAL TRIAL: NCT06434649
Title: Application of the Extra-fascial Robot Assisted Radical Prostatectomy Via the Posterior Approach in Intermediate or High Risk Patients: a Prospective, Multicenter, Double-blind, Randomized Controlled Study
Brief Title: Posterior Extra-fascial RARP in Intermediate or High Risk Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ning Xu (Other)
Collaborators: Fujian Cancer Hospital (Other Government); Zhongshan Hospital Xiamen University (Other); Fuzhou General Hospital (Other); Longyan City First Hospital (Other); The First Hospital of Jilin University (Other); The First Affiliated Hospital of Nanchang University (Other); Ningbo No. 1 Hospital (Other); Hainan People's Hospital (Other); Second Affiliated Hospital of Third Military Medical University (Other); Zhejiang University (Other); Huashan Hospital (Other)
Responsible Party: Sponsor-Investigator, Ning Xu, Head of Urology, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FirstAHFujian-Ning Xu
Record Dates: First submitted 2024-05-10; First posted 2024-05-30 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-09

CONDITIONS: Surgical Procedure, Unspecified; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind technique will be used in this study. The blinding process will be done by a statistician unrelated to this clinical trial. Treatment group assignment will not be known to the subject or to the study followers or to the investigator who clinically evaluates the subject for the entire duration of the trial. Allocation concealment was achieved in this study through an interactive response system. In the absence of serious complications or other emergencies in the subjects during the study period, normal procedures were followed for revealing blinding, this study provides for the use of secondary blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the posterior approach extrafascial technique group (Experimental): In 2010, Italian urologist Dr Bocciardi carried out the first clinical practice of separation and resection of the prostate via the vesicorectal fossa, and this new surgical procedure was called Retzius-sparing Robotic Assisted Radical Prostatectomy (RS-RARP). In recent years, the posterior approach extrafascial technique of RS-RARP which has been used to widely resect the prostate and its surrounding fascia and neurovascular bundles, compared with RS-RARP, has been proposed to provide more complete resection of the tumour and reduce the rate of positive margins. The patients are included into the posterior approach extrafascial technique group who undergo the posterior approach extrafascial technique of RS-RARP.
  Interventions: Procedure: Extrafascial robotic assisted radical prostatectomy via posterior approach
- the anterior approach extrafascial technique group (Active Comparator): Anterior approach extrafascial technique is the most traditional method of radical prostatectomy for prostate cancer, in which the prostate is tied ventrally to expose the prostate by cutting the deep dorsal penile vein complex and the surrounding ligaments and fascia, and intraoperatively extensive resection is required to remove the prostate and its surrounding fascia and neurovascular bundles. The patients are included into the anterior approach extrafascial technique group who undergo the anterior approach extrafascial technique robotic assisted radical prostatectomy.
  Interventions: Procedure: Extrafascial robotic assisted radical prostatectomy via anterior approach

INTERVENTIONS:
Procedure: Extrafascial robotic assisted radical prostatectomy via posterior approach — Extrafascial robotic assisted radical prostatectomy via posterior approach will be applied in the intermediate or high risk patients.
  Arms: the posterior approach extrafascial technique group
Procedure: Extrafascial robotic assisted radical prostatectomy via anterior approach — Extrafascial robotic assisted radical prostatectomy via anterior approach will be applied in the intermediate or high risk patients.
  Arms: the anterior approach extrafascial technique group

SUMMARY:
This study was designed as a prospective, multicentre, double-blind, randomised controlled clinical trial. It aims to investigate the feasibility and safety of the posterior approach extrafascial technique and the anterior approach extrafascial technique in robot-assisted radical prostatectomy (RARP) for intermediate- and high-risk prostate cancer patients, to compare the oncological prognosis, functional prognosis, and safety of the two techniques in intermediate- and high-risk prostate cancer patients, and to provide evidence-based medical evidence for the choice of surgical treatment modality for intermediate- and high-risk prostate cancer patients.

DETAILED DESCRIPTION:
This study was designed as a prospective, multicentre, double-blind, randomised controlled clinical trial. It aims to investigate the feasibility and safety of the posterior approach extrafascial technique and the anterior approach extrafascial technique in robot-assisted radical prostatectomy (RARP) for intermediate- and high-risk prostate cancer patients, to compare the oncological prognosis, functional prognosis, and safety of the two techniques in intermediate- and high-risk prostate cancer patients, and to provide evidence-based medical evidence for the choice of surgical treatment modality for intermediate- and high-risk prostate cancer patients.

About 118 subjects will be enrolled in this study in a total of 12 research centres across the country, and eligible subjects will be randomly assigned to the posterior approach extrafascial technique group and the anterior approach extrafascial technique group in a 1:1 ratio. All subjects routinely underwent comprehensive and systematic physical examination, laboratory tests and imaging examinations before surgery. After surgery, subjects were followed up at 1 week (visit 2, day 14±2), 1 month (visit 3, day 28±5), 3 months (visit 4, day 90±7), 6 months (visit 5, day 180±7), and 12 months (visit 6, day 360±14) after removal of the urinary catheter after the surgery, and then annually thereafter (visit 7), with urine control rate (defined as 0/ 1 pad) and 24-h pad weight questionnaires, PSA examination, International Prostate Symptom Score (IPSS), International Consultation on Incontinence Questionnaire Short Form (ICI-QSF), International Index of Erectile Function (IIEF), and related scores such as General Health-Related Quality of Life (EORTC QLQ-C30) and Prostate Cancer-Specific Quality of Life (QLQ-PR25). ) and other relevant scores; in case of clinical suspicion of local recurrence, imaging (pelvic MRI), whole-body bone imaging in patients with bone pain, and whole-body PET/CT if necessary. Subjects will be monitored and evaluated for adverse events (AE) throughout the trial. Subjects will participate in the clinical trial for an expected duration of approximately 1 year, after which they will be followed up periodically according to the usual follow-up strategy.

ELIGIBILITY:
Inclusion Criteria:

1. intermediate- and high-risk prostate cancer patients assessed by comprehensive clinical evaluation;
2. prostate volume <80 ml;
3. life expectancy of patients >10 years;
4. patients sign the "informed consent";
5. Routine preoperative examination has been improved (chest CT, electrocardiogram, and color Doppler echocardiography), and there is no serious basic disease. After clinical evaluation, it can tolerance robot-assisted radical prostatectomy (RARP).

Exclusion Criteria:

1. life expectancy <10 years;
2. comorbidities with other malignancies;
3. uncorrected coagulation dysfunctions;
4. patients with severe underlying diseases such as severe pulmonary insufficiency who could not tolerate the surgery;
5. patients or family members who did not accept radical prostatectomy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of continence | 1 week after postoperative removal of the urinary catheter
  rate of the preservation of urinary control function at 1 week after postoperative removal of the urinary catheter status
voiding score | through study completion, an average of 1 year
  according to International Consultation on Incontinence Questionnaire Short Form, change in voiding score from baseline period at each visit viewpoint
erectile function score | through study completion, an average of 1 year
  according to International Index of Erectile Function, change in erectile function score from baseline period at each visit viewpoint

SECONDARY OUTCOMES:
the rate of positive specimen margins | after surgery, , an average of 1 year
  the rate of positive specimen margins after surgery
quality of life scores | through study completion, an average of 1 year
  according to EORTC QLQ-C30, quality of life scores at each visit
biochemical recurrence or imaging recurrence/progression | through study completion, an average of 1 year
  biochemical recurrence or imaging recurrence/progression at each visit
overall survival time | From date of randomization until date of death from any cause, an average of 5 year
  deaths (overall survival time) at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Xue-Yi Xue, Study Director — the First Affiliated Hospital, Fujian Medical University
Locations (1):
- first hospital affiliated of Fujian medical university, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No